CLINICAL TRIAL: NCT07049276
Title: Randomized Controlled Trial of Selective Index Lymph Node Resection Versus Therapeutic Lymph Node Dissection After Neoadjuvant Immunotherapy for Stage IIIB-D Melanoma
Brief Title: The Multicentre Selective Lymphadenectomy Trial - 3
Acronym: MSLT-3
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Melanoma Institute Australia (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: MIA2024/501
Record Dates: First submitted 2025-05-24; First posted 2025-07-03 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Cutaneous Melanoma, Stage III
Keywords: Neoadjuvant; Non-inferiority; Randomised controlled trial; Adverse events; Quality of life; Healthcare economics; Index lymph node resection; Therapeutic lymph node dissection; Surgical morbidity
MeSH Terms: conditions — Melanoma

STUDY DESIGN:
Intervention Model Description: Non-inferiority
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Index Lymph Node (Experimental): The largest affected (index) lymph node marked with a clip under ultrasound or X-ray guidance and then removed after neoadjuvant therapy for the pathological response to be determined. The response then dictates the next step of management
  Interventions: Procedure: Index lymph node resection
- Therapeutic lymph node dissection (Active Comparator): Complete removal of all nodes in the regional lymph node basin
  Interventions: Procedure: Therapeutic lymph node dissection

INTERVENTIONS:
Procedure: Index lymph node resection — The largest lymph node affected with melanoma
  Arms: Index Lymph Node
Procedure: Therapeutic lymph node dissection — Removal of all nodes in the melanoma affected lymph node basin
  Arms: Therapeutic lymph node dissection

SUMMARY:
The goal of this clinical trial is to demonstrate that there is no difference (non-inferiorty) in the 2 year recurrence-free survival (RFS) between 2 different surgical approaches for clinical Stage III melanoma. Following 6 weeks of standard neaodjuvant immunotherapy, patients will undergo either selective index lymph node resection (ILN) (identified at baseline as the largest affected lymph node) or the standard of care therapeutic lymph node dissection (TLND). The secondary aims are to assess if patients who are managed without TLND will have a reduction in surgical complications (less wound problems & lymphoedema), an improved quality of life, at a lower healthcare utilisation.

DETAILED DESCRIPTION:
The standard treatment under current guidelines for patients who have melanoma that has spread to the lymph nodes (Stage III disease) is a 'therapeutic lymph node dissection' or 'TLND'. This is the removal of all of the lymph nodes in the affected area, such as in the armpit, neck or groin. TLND surgery

Several clinical trials over the past 10 to 15 years have shown that treatment with immune system boosting drugs (known as immunotherapy) can help the body to better identify and attack the tumour cells. This is now used routinely for tumour that has spready beyond the lymph nodes (Stage IV disease) in melanoma and many other cancers.

When immunotherapy is given before TLND surgery (known as neoadjuvant therapy) the body can launch an increased immune response against the tumour cells to reduce or remove the amount of tumour before surgery. Neoadjuvant therapy for melanoma is typically given over 6 weeks before surgery. Patients may have further drug therapy and /or radiotherapy after TLND surgery to minimise the risk of recurrence.

At surgery after neoadjuvant immunotherapy, the removed lymph node tissue is examined by a pathologist who will then classify the amount of tumour cells left in the lymph nodes. Recent clinical trials have shown that 46-70% of patients have less than 10% of melanoma cells left in the lymph nodes. This is called a 'major pathological response' or 'MPR'. After 5 years, approximately 70% of patients having an MPR do not have a recurrence of melanoma. Neoadjuvant immunotherapy is now standard care for Stage III melanoma in Australia and other countries.

Both immunotherapy and TLND surgery have side effects. Some of these are of short duration and some last many months. Some of the side effects from immunotherapy include general nausea, diarrhoea, skin rash but also diabetes, thyroid or liver problems. Surgery may result in some pain, wound infection, wound breakdown, or short and long term lymphoedema - where fluid doesn't drain properly from the arms or legs, depending on where the original lymph node surgery was done.

A recent small clinical trial of 99 patients tested if patients who have neoadjuvant therapy can omit the need for TLND surgery, without changing the risk of recurrence. Patients in this study had the largest affected (index) lymph node marked with a clip under ultrasound or X-ray guidance before neoadjuvant therapy. After 6 weeks of neoadjuvant immunotherapy, the index lymph node was removed in a minor operation and the pathological response classified. Sixty-one percent of patients had an MPR and did not have any further surgery. After 2 years, 93% of these patients did not have a recurrence of melanoma. Patients without an MPR had TLND surgery and between 63 and 75% had no recurrence by 2 years.

This recent trial was too small to provide sufficient evidence for a change in standard treatment after neoadjuvant immunotherapy for patients having an MPR. We therefore plan to conduct a trial that is large enough to test if the new approach of index lymph node resection is not worse than the current standard care with TLND as measured by the number of people without melanoma recurrence within 2 years. This type of trial is known as a 'non-inferiority' trial. If index node resection is no worse than TLND, we also need to assess if there is a difference in the side effects or each type of surgery and in the quality of life experienced by patients. We also need to examine if there is any difference in the costs to patients and to the healthcare system for either surgery and the long term outcomes.

This is a randomised trial which means people are put into one of two groups by chance (randomly, or like tossing a coin). For patients who have an MPR to neoadjuvant therapy, half will have index lymph node removal with no further surgery and half the current standard of TLND surgery. Patients who do not have an MPR will have the standard TLND. All patients will have regular appointments with their surgeon to check for signs if the melanoma has returned and the study team will follow progress for up to 10 years.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female patients ≥ 18 years of age at the time of consent
2. Written informed consent
3. Cytologically or histologically confirmed, resectable pathological Stage IIIB, C or D (Any T, N1b, N2b, N2c, N3b, or N3c) cutaneous or unknown primary melanoma, with or without primary tumour in situ
4. A minimum of one macroscopic lymph node, defined as:

   * A palpable node, confirmed by pathology
   * A non-palpable node, but enlarged per RECIST 1.1 criteria (≥ 15 mm in shortest diameter) and confirmed by pathology
   * An ultrasound or PET/CT scan positive lymph node of any size, confirmed by pathology.
5. Up to 3 satellite (defined as any foci of clinically evident cutaneous and/or subcutaneous metastases occurring within 2 cm of but discontinuous from the primary melanoma) or in-transit metastases (defined as clinically evident cutaneous and/or subcutaneous metastases occurring >2 cm from the primary melanoma in the region between the primary and the regional lymph node basin) are permitted if they are completely resectable.
6. Lymph node involvement in the groin (iliac, inguinal or both), axilla or neck only and may be unilateral or bilateral. Concurrent popliteal, epitrochlear or triangular intermuscular space (TIS) nodes permitted, as long as fully resectable.
7. Tumour amenable to a newly obtained core biopsy of a lesion which has not been previously irradiated. Archival tissue from a past primary or nodal lesion (if applicable) or tissue taken for current diagnosis will also be collected if available.
8. Systemic neoadjuvant immunotherapy is scheduled for administration with at least one PD-(L)-1 check point inhibitor (e.g. nivolumab, pembrolizumab, cemiplimab). The immunotherapy regimen may include other checkpoint inhibitors (e.g. ipilimumab, relatlimab, fianlimab). The patient should meet the fitness for treatment requirements as detailed in the relevant regulatory-approved Product Information or Summary of Product Characteristics.
9. Neoadjuvant course of treatment to be no longer than 6 weeks (allows for a maximum of 3 cycles at weeks 0, 3 and 6).
10. Eastern Cooperative Oncology Group (ECOG) performance status of 0-1.
11. Anticipated life expectancy of > 5 years.

Exclusion Criteria:

1. Uveal or mucosal melanoma.
2. Isolated satellite or in-transit metastases only (without any cytological or histological proven lymph node involvement).
3. Involvement of any lymph node basin other than groin, axilla or neck. Concurrent popliteal, epitrochlear or triangular intermuscular space (TIS) nodes permitted, as long as fully resectable.
4. Clinical or radiographic evidence of distant metastasis (any AJCC 8th ed M Stage).
5. Previous history of lymph node surgery to the same nodal basin, that was more extensive than a sentinel lymph node biopsy (SLNB).
6. Previous radiotherapy to the same nodal basin.
7. Any contraindication to the administration of nivolumab, ipilimumab, pembrolizumab or relatlimab per regulatory-approved product information and / or medical oncologist.
8. Prior anti-PD-1, CTLA-4, PDL-1 or LAG 3 antibody exposure, or an agent directed to another stimulatory or co-inhibitory T-cell receptor for any disease or any chemotherapy or experimental local or systemic drug treatment.
9. A plan to administer targeted therapy or any non-checkpoint inhibitor immunotherapy, or any intralesional therapy for melanoma in the neoadjuvant setting.
10. A plan to administer any experimental immunotherapy as part of a clinical trial in the neoadjuvant setting.
11. Known additional malignancies (unless adequately treated) active within the previous 3 years, except for locally curable cancers that have been apparently cured. The following malignancies, if undergone successful definitive resection or curative treatment, are permitted:

    * Basal cell carcinoma of the skin
    * Squamous cell carcinoma of the skin
    * Carcinoma in situ (e.g. breast carcinoma, cervical cancer in situ, but excluding carcinoma in situ of the bladder) that have undergone potentially curative therapy
    * Prostatic intraepithelial neoplasia
    * In situ melanoma
    * Atypical melanocytic hyperplasia
    * Stage I melanoma
    * Other malignancies for which the patient has been disease free for 3 years, not requiring active anti-cancer therapy.
12. An active autoimmune disease or a requirement for chronic systemic steroid therapy (in dosing exceeding 10 mg daily of prednisone equivalent) or any other form of immunosuppressive therapy within 14 days prior to the first dose of study treatment. The following are permitted:

    * Replacement therapy (e.g. thyroxine, insulin, or physiologic corticosteroid replacement therapy for adrenal or pituitary insufficiency, etc)
    * Inhaled or intranasal corticosteroids (with minimal systemic absorption) may be continued if patient is on a stable dose
    * Non-absorbed intra-articular steroid injections.
13. Has had an allogenic tissue/solid organ transplant.
14. Active Hepatitis B (defined as Hepatitis B surface antigen [HBsAg] reactive) or Hepatitis C virus (defined as HCV RNA [qualitative] is detected) infection. Note: no testing for Hepatitis B and Hepatitis C is required unless mandated by local health authority.
15. Has a known history of Human Immunodeficiency Virus (HIV). Note: no testing for HIV is required unless mandated by local health authority.
16. Pregnant or breastfeeding females.
17. Concurrent medical or social conditions that may prevent the patient from attending assessments or procedures per schedule.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1500 (Estimated)
Dates: Start 2025-10-01 (Actual); Primary Completion 2030-08 (Estimated); Study Completion 2040-08 (Estimated)

PRIMARY OUTCOMES:
Recurrence free survival | 2 years
  The proportion of patients with a major pathological response alive and disease-free from the time of surgery to the end of 2 years follow up

SECONDARY OUTCOMES:
The rate of escalation to a therapeutic lymph node dissection (TLND) in the ILN arm due to isolated nodal recurrence in the ILN nodal basin | 2 years
  Proportion of patients with a major pathological response (complete pathological response or near complete pathological response) in the index lymph node arm who have disease recurrence involving the same lymph node basin requiring complete dissection
The salvage rate with surgery, radiotherapy or new systemic therapy post operatively for disease recurrence in each surgical arm with a major pathological response (complete pathological response or near complete pathological response) | 2 years
  Proportion of patients requiring any additional treatment for any disease recurrence following a complete or near complete pathological response
Distant metastasis free-survival | 2 years
  Proportion of patients with distant metastases from randomisation to the date of first distant metastases diagnosis in each surgical arm, following a major pathological response (complete pathological response or near complete pathological response)
Overall survival | 10 years
  Proportion of patients who die, from the date of randomisation to the date of death from any cause
Surgery-related adverse events | 2 years
  Surgical related adverse events using CTCAE version 5.0
Surgery-related adverse events | 3 weeks, 12 weeks and 48 weeks post surgery
  Surgical related adverse events using Clavien-Dindo scale
Patient-rated quality of life QLQ C30 | 6, 12, 24, 36 and 48 weeks
  Baseline EUROQOL QLQ-C30,scores compared to scores reported over the duration on study
Patient-rated quality of life EQ 5D5L | 6, 12, 24, 36 and 48 weeks
  Baseline EQ-5D-5L compared to scores reported over the duration on study
Patient-rated quality of life FACT-M | 6, 12, 24, 36 and 48 weeks
  Week 6 FACT-M scores compared to scores reported over the duration on study
Concordance of metabolic response with pathological response | week 6
  The PET results correlated with the pathological response
Concordance of metabiolic response with RECIST response | week 6
  The PET results correlated with the CT response
Concordance of metabolic response with circulating ctDNA | week 6
  The PET results correlated with the volume of circulating tumour DNA in the blood
Health-related economic costs | 2 years
  Comparison of the health-related costs related to each surgical procedure and its outcomes

OTHER OUTCOMES:
To identify prognostic and predictive biomarkers for recurrence | 2 years
  Comparison of multi-omic biomarkers from baseline with clinical outcomes

CONTACTS AND LOCATIONS:
Overall Officials: Alexander CJ van Akkooi, Study Chair — Melanoma Institute Australia
Locations (6):
- Cedars-Sinai Medical Centre, Los Angeles, California, United States
- Melanoma Institute Australia, Wollstonecraft, New South Wales, Australia
- Sunnybrook Health Sciences Centre, Toronto, Ontario, Canada
- San Maria della Misericordia Hospital, Perugia, Italy
- North Shore Hospital, Takapuna, Auklnad, New Zealand
- The Royal Marsden, London, United Kingdom